CLINICAL TRIAL: NCT01198509
Title: Role of Oral and Intestinal Microbiota in Rheumatoid Arthritis (RA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 09-0658; RC2AR058986 (NIH)
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Periodontal Disease
Keywords: rheumatoid arthritis; psoriatic arthritis; periodontitis; microbiota; microbiome; vancomycin; doxycycline; T cell; Th17
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Periodontal Diseases; Periodontitis | interventions — Doxycycline; Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rheumatoid Arthritis (RA) - doxycycline (Active Comparator): Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive doxycycline, 100 mg twice a day, for 2 months.
  Interventions: Drug: doxycycline
- Rheumatoid Arthritis (RA) - vancomycin (Active Comparator): Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive vancomycin, 250 mg four times a day, for 2 weeks
  Interventions: Drug: vancomycin
- RA, PsA, healthy (No Intervention): Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive no antibiotic treatment for comparison with Doxycycline- and Vancomycin-treated patients.
  Patients with psoriatic arthritis (PsA), to provide baseline samples of oral and intestinal microbiota for comparison with RA patients.
  Healthy individuals with no history of arthritis, to provide baseline samples of oral and intestinal microbiota for comparison with RA patients.

INTERVENTIONS:
Drug: doxycycline — doxycycline - 100 mg twice per day, for 2 months
  Other Names: Vibramycin
  Arms: Rheumatoid Arthritis (RA) - doxycycline
Drug: vancomycin — vancomycin, 250 mg four times a day, for 2 weeks
  Other Names: Vancocin
  Arms: Rheumatoid Arthritis (RA) - vancomycin

SUMMARY:
Rheumatoid arthritis (RA) is an inflammatory form of arthritis that causes joint pain and damage. RA attacks the lining of the joints (synovium), causing swelling that can result in aching and throbbing, and eventually deformity. Even though there have been many advances in the treatment of RA, psoriatic arthritis (PsA), and other inflammatory arthritis, doctors still do not know what causes this inflammation in joints. It is likely that RA occurs as a result of a complex combination of factors, including a person's genes; lifestyle choices, such as smoking and diet; and things in a person's environment, including bacteria or viruses. This study investigates the hypothesis that bacteria living in a person's mouth and/or intestinal tract are responsible, at least in part, for the development of Rheumatoid Arthritis. The investigators believe that by killing those bacteria with antibiotics, they might be able to understand how the immune system works and, maybe, what causes RA.

DETAILED DESCRIPTION:
If you would like to participate in this study, we will first ask you several questions regarding the status of your arthritis, the medications you use or have used in the recent past, your social and dietary habits, and your medical and surgical history. If your answers tell us that you are the right patient for our study, we will go over a consent form which describes in more detail how we will study your intestinal and mouth bacteria, the immune cells in your blood and other genes, enzymes and proteins that tell us about your disease status.

If you have Psoriatic Arthritis (PsA) or are healthy with no history of arthritis, and would like to participate in this study, your participation would involve only one or two visits, and no treatment.

If you have Rheumatoid Arthritis (RA), your participation would involve six visits, and you would be randomly assigned to receive treatment with the antibiotic doxycycline, or the antibiotic vancomycin, or no antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis (RA) patients must meet American College of Rheumatology (ACR) criteria for RA
* RA patients: duration of disease will be greater than 6 weeks and less than 2 years.
* RA patients should have a Disease Activity Score 28 (DAS28) greater than or equal to 5.
* PsA patients will be required to have disease duration and DAS28 similar to the RA patients, and to meet Moll and Wright criteria for PsA.
* Allowable medications for both groups at study entry will include: prednisone (or equivalent) 5 mg or less per day (stable dose for at least 2 months); methotrexate 15 mg or less per week (stable dose for at least 2 months); and nonsteroidal anti-inflammatory drugs (NSAIDs) at FDA-approved doses.
* Healthy controls will be age- and sex-matched individuals with no personal or family history of inflammatory arthritis.

Exclusion Criteria:

* Patients who are unable to provide informed consent.
* Pregnant or lactating women.
* Recent (<3 months prior) use of any antibiotic therapy
* Current consumption of probiotics
* Current extreme diet (parenteral nutrition, macrobiotic diet, etc.)
* Prednisone >5 mg/day or equivalent
* Use of other disease-modifying antirheumatic drugs (DMARDs) with known antibiotic properties (Gold salts, hydroxychloroquine, sulfasalazine or minocycline).
* Use of biologic DMARDs
* Known inflammatory bowel disease
* Known gastrointestinal (GI) tract neoplasm.
* Recent GI tract infection (gastroenteritis, colitis, diverticulitis, appendicitis)
* Chronic unexplained diarrhea.
* Any GI tract surgery leaving permanent residua (e.g., gastrectomy; bariatric surgery; colectomy)
* Significant liver, renal or peptic ulcer disease, defined as:

  * Liver: aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 x upper limit of normal (ULN)
  * Renal: Creatinine >1.5 or endstage renal disease
  * Peptic ulcer disease: recent ulcer or GI bleed (within past 12 months)
* Inability or unwillingness to abstain from alcohol consumption.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven B. Abramson, MD, Principal Investigator — NYU Langone Health; Jose U. Scher, MD, Study Director — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Hospital for Joint Diseases, New York, New York
  - Bellevue Hospital, New York, New York

REFERENCES:
- [Background] Scher JU, Abramson SB. The microbiome and rheumatoid arthritis. Nat Rev Rheumatol. 2011 Aug 23;7(10):569-78. doi: 10.1038/nrrheum.2011.121. PMID 21862983
- [Background] Honda K, Littman DR. The microbiome in infectious disease and inflammation. Annu Rev Immunol. 2012;30:759-95. doi: 10.1146/annurev-immunol-020711-074937. Epub 2012 Jan 6. PMID 22224764
- [Background] Littman DR, Pamer EG. Role of the commensal microbiota in normal and pathogenic host immune responses. Cell Host Microbe. 2011 Oct 20;10(4):311-23. doi: 10.1016/j.chom.2011.10.004. PMID 22018232
- [Background] Brusca SB, Abramson SB, Scher JU. Microbiome and mucosal inflammation as extra-articular triggers for rheumatoid arthritis and autoimmunity. Curr Opin Rheumatol. 2014 Jan;26(1):101-7. doi: 10.1097/BOR.0000000000000008. PMID 24247114
- [Background] Scher JU, Abramson SB. Periodontal disease, Porphyromonas gingivalis, and rheumatoid arthritis: what triggers autoimmunity and clinical disease? Arthritis Res Ther. 2013;15(5):122. doi: 10.1186/ar4360. PMID 24229458
- [Result] Scher JU, Ubeda C, Equinda M, Khanin R, Buischi Y, Viale A, Lipuma L, Attur M, Pillinger MH, Weissmann G, Littman DR, Pamer EG, Bretz WA, Abramson SB. Periodontal disease and the oral microbiota in new-onset rheumatoid arthritis. Arthritis Rheum. 2012 Oct;64(10):3083-94. doi: 10.1002/art.34539. PMID 22576262
- [Result] Tang W, Lu Y, Tian QY, Zhang Y, Guo FJ, Liu GY, Syed NM, Lai Y, Lin EA, Kong L, Su J, Yin F, Ding AH, Zanin-Zhorov A, Dustin ML, Tao J, Craft J, Yin Z, Feng JQ, Abramson SB, Yu XP, Liu CJ. The growth factor progranulin binds to TNF receptors and is therapeutic against inflammatory arthritis in mice. Science. 2011 Apr 22;332(6028):478-84. doi: 10.1126/science.1199214. Epub 2011 Mar 10. PMID 21393509
- [Result] Scher JU, Sczesnak A, Longman RS, Segata N, Ubeda C, Bielski C, Rostron T, Cerundolo V, Pamer EG, Abramson SB, Huttenhower C, Littman DR. Expansion of intestinal Prevotella copri correlates with enhanced susceptibility to arthritis. Elife. 2013 Nov 5;2:e01202. doi: 10.7554/eLife.01202. PMID 24192039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: January 2010 - August 2012 Locations: Medical clinics and faculty practice offices
Groups:
- Rheumatoid Arthritis (RA) - Doxycycline: Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive doxycycline, 100 mg twice a day, for 2 months.
  doxycycline: doxycycline - 100 mg twice per day, for 2 months
  N=5 (actual)
- Rheumatoid Arthritis (RA) - Vancomycin: Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive vancomycin, 250 mg four times a day, for 2 weeks
  vancomycin: vancomycin, 250 mg four times a day, for 2 weeks
  N=10 (actual)
- Rheumatoid Arthritis (RA) Randomized to no Treatment: Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive no antibiotic treatment for comparison with Doxycycline- and Vancomycin-treated patients.
  N=19 (actual)
- Early RA Cross-sectional Cohort: Patients with rheumatoid arthritis (RA) meeting inclusion criteria who opted to participate ONLY in cross-sectional analysis (one-time sample collection equivalent to the involvement of PsA and health control subjects).
  N=66 (actual)
- Psoriatic Arthritis (PsA): Patients with psoriatic arthritis (PsA), to provide baseline samples of oral and intestinal microbiota for comparison with RA patients.
  N=20 (actual)
- Healthy Volunteers: Healthy individuals with no history of arthritis, to provide baseline samples of oral and intestinal microbiota for comparison with RA patients.
  N=58 (actual)
Period: Overall Study
Arm/Group | Rheumatoid Arthritis (RA) - Doxycycline | Rheumatoid Arthritis (RA) - Vancomycin | Rheumatoid Arthritis (RA) Randomized to no Treatment | Early RA Cross-sectional Cohort | Psoriatic Arthritis (PsA) | Healthy Volunteers
Started | 5 | 10 | 19 | 66 | 20 | 58
Completed | 4 (Patient declined further participation after enrollment and allocation to treatment group) | 10 | 19 | 66 | 20 | 58
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rheumatoid Arthritis (RA) Randomized to no Treatment: Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive no antibiotic treatment and followed prospectively for 6 months, for comparison with Doxycycline- and Vancomycin-treated patients.
- Early RA Cross-sectional Cohort: Patients with rheumatoid arthritis (RA) meeting inclusion criteria who opted to participate ONLY in cross-sectional analysis (one-time sample collection equivalent to the involvement of PsA and health control subjects).
- Psoriatic Arthritis (PsA): Patients with psoriatic arthritis (PsA), to provide baseline samples of oral and intestinal microbiota for comparison with RA patients.
- Healthy Volunteers: Healthy individuals with no history of arthritis, to provide baseline samples of oral and intestinal microbiota for comparison with RA patients.
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis (RA) - Doxycycline | Rheumatoid Arthritis (RA) - Vancomycin | Rheumatoid Arthritis (RA) Randomized to no Treatment | Early RA Cross-sectional Cohort | Psoriatic Arthritis (PsA) | Healthy Volunteers | Total
Number analyzed (Participants) | 5 | 10 | 19 | 66 | 20 | 58 | 178
Age, Continuous [Mean (Full Range); unit: years] | 44.0 [31 to 68] | 41.5 [24 to 63] | 39.2 [26 to 69] | 49.1 [20 to 85] | 45.5 [26 to 73] | 40.7 [21 to 62] | 44.2 [20 to 85]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 10 | 18 | 58 | 19 | 58 | 167
  >=65 years | 1 | 0 | 1 | 8 | 1 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 14 | 53 | 11 | 50 | 139
  Male | 1 | 3 | 5 | 13 | 9 | 8 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4 | 5 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 17 | 1 | 9 | 31
  White | 1 | 2 | 1 | 16 | 6 | 12 | 38
  More than one race | 2 | 6 | 14 | 29 | 8 | 35 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 15 | 41 | 8 | 43 | 117
  Not Hispanic or Latino | 2 | 3 | 4 | 25 | 12 | 15 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 19 | 66 | 20 | 58 | 178

OUTCOME MEASURES:

1. Primary Outcome: Alteration of Microbiota, Alteration of T Cell Function/Activation
Description: Oral and intestinal microbiota, and T cell function and activation, will be assessed at baseline, and at 1, 2, 3, 4 and 5 months after baseline, to determine whether changes are associated with vancomycin treatment versus doxycycline treatment versus no treatment.
  Results are reported as number of participants who experienced changes in oral/intestinal microbiota, T cell function/activation.
  Methods/criteria to assess change in microbiota: change in relative abundance of microorganisms at genus and species level (as assessed high-throughput 16S rDNA sequencing).
  Methods/criteria to assess change in T cell function/activation: change in percentage of inhibition of regulatory T cells as measured by interferon gamma levels in in-vitro assays.
Time Frame: 6 months
Population: Primary outcome only evaluated in first three groups of RA patients: 4 randomized to treatment with doxycycline; 10 randomized to treatment with vancomycin; 19 randomized to no treatment.
Measure: Number; unit: participants
Groups:
- Rheumatoid Arthritis (RA) Randomized to no Treatment: Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive no antibiotic treatment, followed prospectively for 6 months, for comparison with Doxycycline- and Vancomycin-treated patients.
  N=19 (actual)
Arm/Group | Rheumatoid Arthritis (RA) - Doxycycline | Rheumatoid Arthritis (RA) - Vancomycin | Rheumatoid Arthritis (RA) Randomized to no Treatment | Early RA Cross-sectional Cohort | Psoriatic Arthritis (PsA) | Healthy Volunteers
Number analyzed (Participants) | 4 | 10 | 19 | 66 | 20 | 58
participants
  Change in oral/intestinal microbiota | 4 | 10 | 2 | 0 | 0 | 0
  Change in T cell function/activation | 2 | 6 | 19 | 0 | 0 | 0

2. Secondary Outcome: Mean Units Change in DAS28 From Baseline to 6 Months
Description: DAS28 (disease activity score with 28 joint count). Possible score range: 0 to 10. This is a composite index calculated from 4 measures: two from a physician (28 tender joint count, 28 swollen joint count), one from the patient (patient global estimate of disease activity), and one laboratory biomarker (erythrocyte sedimentation rate or ESR). A score of 0 represents best possible health status (no apparent disease activity) and 10 represents worst possible.
  The outcome is reported as mean change in DAS28 score from baseline to 6 months. The mean changes reported are negative values for downward change in score (i.e., improvement in health status).
Time Frame: 6 months
Population: Please note that only the first 3 groups (RA doxycycline, RA vancomycin, and RA randomized to no treatment) were analyzed for change from baseline to six months (outcomes). Groups 4, 5 and 6 (RA cross-sectional, Psoriatic Arthritis, and Healthy Volunteers) were analyzed for baseline measures only in a cross-sectional comparison.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Rheumatoid Arthritis (RA) Randomized to no Treatment: Patients with rheumatoid arthritis (RA) meeting inclusion criteria, randomized to receive no antibiotic treatment and followed prospectively for 6 months, for comparison with Doxycycline- and Vancomycin-treated patients.
  N=19 (actual)
Arm/Group | Rheumatoid Arthritis (RA) - Doxycycline | Rheumatoid Arthritis (RA) - Vancomycin | Rheumatoid Arthritis (RA) Randomized to no Treatment | Early RA Cross-sectional Cohort | Psoriatic Arthritis (PsA) | Healthy Volunteers
Number analyzed (Participants) | 4 | 10 | 19 | 0 | 0 | 0
units on a scale | -1.3 [-1.7 to -0.4] | -1.5 [-4.4 to -0.2] | -2.5 [-3.9 to -0.9] |  |  |

ADVERSE EVENTS:
Time Frame: Duration of the study, up to 6 months
Arm/Group | Rheumatoid Arthritis (RA) - Doxycycline | Rheumatoid Arthritis (RA) - Vancomycin | RA, PsA, Healthy
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10 | 0/163
Other Adverse Events (participants affected / at risk) | 0/4 | 1/10 | 0/163
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rheumatoid Arthritis (RA) - Doxycycline (N=4) | Rheumatoid Arthritis (RA) - Vancomycin (N=10) | RA, PsA, Healthy (N=163)
stomach pain/loose stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Resolved within 24 hours. Possibly related to study treatment. Participant continued treatment and completed study.

LIMITATIONS AND CAVEATS:
Interpretation of results is limited by very small sample size. It should be noted that this was intended as a proof-of-concept study, and not a fully-powered clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No